CLINICAL TRIAL: NCT04642443
Title: A Prospective, Two-Stage, Non-randomized, Multi-center Within Patient Comparison Study to Evaluate the SENSE Device's Ability to Detect Intracranial Hemorrhage
Brief Title: Evaluate the SENSE Device's Ability to Monitor and Detect Intracranial Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sense Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SENSE-003
Record Dates: First submitted 2020-11-19; First posted 2020-11-24 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Intracranial Hemorrhages; Traumatic Brain Injury
MeSH Terms: conditions — Intracranial Hemorrhages; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intracranial Hemorrhage (Active Comparator): The SENSE device transmits a low power tailored electro-magnetic (EM) pulse in the radio-frequency range across the patient's brain and detects changes in the signal that may indicate intracranial hemorrhage. The device consists of three parts:
  1. A molded plastic headpiece containing the antenna array
  2. An intermediate control unit that contains:
     a. The driving electronics for the array of antennae
  3. A processing control unit that contains:
     1. A spectrum analyzer
     2. The operating software that controls the device function and data acquisition, processing and archiving.
     3. The user interface for inputting patient information and displaying the output of the data
  Interventions: Device: SENSE Device
- Traumatic Brain Injury (Active Comparator): The SENSE device transmits a low power tailored electro-magnetic (EM) pulse in the radio-frequency range across the patient's brain and detects changes in the signal that may indicate intracranial hemorrhage. The device consists of three parts:
  1. A molded plastic headpiece containing the antenna array
  2. An intermediate control unit that contains:
     a. The driving electronics for the array of antennae
  3. A processing control unit that contains:
     1. A spectrum analyzer
     2. The operating software that controls the device function and data acquisition, processing and archiving.
     3. The user interface for inputting patient information and displaying the output of the data
  Interventions: Device: SENSE Device

INTERVENTIONS:
Device: SENSE Device — The SENSE Device is indicated for the monitoring of intracranial hemorrhage by detecting a suspected increase in blood volume within the cranial vault. It is an adjunctive device to the clinical evaluation in the acute hospital setting of patients 22 years of age or older with suspected or known intracranial hemorrhage. The device is indicated for use to monitor patients for intracranial hemorrhage expansion between CT scans but should not serve as a substitute for these scans.

SUMMARY:
This study is a two-stage, pivotal, prospective, non-randomized, multi-center, within patient comparison of the SENSE device and the standard diagnostic test, head CT scan in patients with a diagnosis of primary spontaneous ICH or traumatic intracranial bleeding for the detection and monitoring of intracranial hemorrhages.

DETAILED DESCRIPTION:
This study is a two-stage, pivotal, prospective, nonrandomized, multi-center, within patient comparison of the SENSE device and the standard diagnostic test, head CT scans. All subjects who meet eligibility criteria should be enrolled. An algorithm has been developed for detecting ICH, which will now be tested in this independent cohort of subjects. CT scans will be grouped into: 1) ICH, or 2) non- ICH. Enrollment will continue until 120 subjects with and 120 without ICH have been enrolled. An interim analysis will occur after ~60 subjects each with and without ICH have been enrolled and the sample size may be increased at the direction of the DMC as warranted. In Stage 1, 150 subjects (with primary spontaneous ICH or traumatic intracranial hemorrhage) were enrolled for the development of a hemorrhage detection algorithm. In Stage 2, the algorithm developed in Stage 1 will be tested in an independent cohort of up to 300 subjects. All subjects who meet eligibility criteria should be enrolled. The gold standard will be the CT results. The algorithm established in Stage 1 will be tested in this independent cohort of subjects. CT scans will be grouped into: 1) ICH or, 2) non-ICH. Enrollment will continue until ~60 subjects each with and without ICH have been enrolled. An interim analysis will occur after ~60 subjects each with and without ICH have been enrolled and the sample size may be increased at the direction of the DMC as warranted. All subjects' CT images will be reviewed by an independent neuroradiology core for classification as ICH or non-ICH, and ICH volume estimation. The treating clinicians and independent neuroradiologist will be blinded to the SENSE device findings.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age 22 years and older
* CT obtained in the mobile stroke unit, emergency department (ED) or hospital

Exclusion Criteria:

* Female patients who are pregnant or lactating
* SENSE device cannot be applied within 6 hours of a standard of care CT,
* Metallic intracranial clip, coil, device (such as ICP monitor), or penetrating metallic shrapnel,
* Metallic EEG leads in place at the time of planned enrollment,
* Open skull fracture (closed skull fracture is not an exclusion),
* Placement of an intraventricular catheter prior to enrollment, Hemorrhagic transformation of ischemic stroke,) as etiology of ICH,
* Treatment with intravenous thrombolysis or embolectomy prior to enrollment,
* Clinical uncertainty about whether intracranial hemorrhage is present on the pre-enrollment head CT, and
* Presence or history of any other condition or finding that, in the investigator's opinion, makes the patient unsuitable as a candidate for SENSE device monitoring or study participation or may confound the outcome of the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 24-hours
  Detection of ICH is the primary endpoint for this study. To establish the sensitivity (primary) and specificity (key secondary) for ICH detection. The results from the CT (ICH versus no ICH) scan will serve as the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Ratcliff, MD, Principal Investigator — Emory University
Locations (1):
- Grady, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No